CLINICAL TRIAL: NCT03067493
Title: Radiofrequency Ablation or Surgical Resection Combined With Neo-MASCT for Primary Hepatocellular Carcinoma: a Randomised, Multicentre Phase II Trial
Brief Title: RFA or Surgical Resection Combined With Neo-MASCT for Primary HCC: a Phase II Trial
Acronym: RAMEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCC008
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Primary Liver Cancer; Radiofrequency Ablation; Immunotherapy; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neo-MASCT group (Experimental): Patients in the treatment group will receive a total of 6 courses of Neo-MASCT treatment. The whole period of Neo-MASCT treatment for each patient will be up to 24 months.Three stratification factors are considered, i.e.tumor size (2.1-3.0cm, 3.1-5.0cm), tumor number (1, >1) and type of surgery (RFA，hepatectomy).
  Interventions: Biological: Neo-MASCT
- Control group (No Intervention): Patients in the control group will be actively monitored during the trial period. Patients will receive assessment every 3 months in the first 3 years.

INTERVENTIONS:
Biological: Neo-MASCT — Patients assigned to Neo-MASCT treatment will receive 18 cycles of neo-MASCT (6 courses), with one cycle every month for the first year and one cycle every 2 months for the second year. Each cycle includes one DCs subcutaneous injection and one CTLs infusion.
  Arms: Neo-MASCT group

SUMMARY:
RAMEC is a phase II, multi-center, randomized trial with a safety test. There will be a safety test to establish the safety and tolerability of Neo-MASCT treatment and assess the immune response to the treatment.The randomized trial will assess DFS and immune response.

DETAILED DESCRIPTION:
The safety test will recruit 10 patients. Following registration they will receive 3 cycles of Neo-MASCT treatment. Patients will be seen at week 1, week 2 and week 4 of every cycle.

Following the safety test, 98 patients will be randomized to the trial across 3 recruiting centers. All patients on the treatment arm will complete up to 18 cycles of Neo-MASCT treatment. Patients on the control arm will be actively monitored after randomization. Blood samples for immune response test will be taken at baseline, cycle 1day 1 and then 3 monthly on day 1 of the subsequent cycles. The planned treatment duration will be until relapse of disease, unacceptable toxicity or withdrawal of consent. The end of the trial will be 24 months after the recruitment of the last patient.

ELIGIBILITY:
Inclusion Criteria before resection/RFA:

1. Aged ≥ 18 years;
2. Primary HCC received RFA/Hepatectomy as the initial treatment; a solitary tumour 2.0-5.0m in diameter; or 2-3 tumours with the largest ≤5.0cm; all without vascular invasion, lymphatic metastasis or distant metastasis (see Appendix 1 for diagnosis criteria).
3. ECOG 0/1 (Appendix 3);
4. Child-Pugh score 5-7 (Appendix 4);
5. A life expectancy of 6 months or more；
6. Adequate haematological, liver and renal function Neutrophil count ≥1.5 x 109/L; platelet count> 60 x 109/L; Haemoglobin concentration≥9.0 g/dL; Serum albumin≥ 3.0 g/dL; A total bilirubin of less than 1.5 times upper limit of normal; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 3 times upper limit of normal; Prothrombin time ≤3s above the control Serum creatinine concentration of 1.5 times the upper limit of the normal range or less; CCR ≥60ml/min
7. Written informed consent

Exclusion Criteria:

1. Pregnant women, lactating women or women planning to be pregnant in 2 years;
2. Intrahepatic metastasis, tumour thrombosis in main trunk or main branches of portal vein, tumour thrombosis in hepatic vein;
3. Systematic use of potent immunosuppressive agents within 6 months or long-term use of them such as corticosteroids, cyclosporine A, et al;
4. Concomitant HIV or HCV infection;
5. Concomitant immunodeficiency diseases or autoimmune diseases (eg. rheumatoid arthritis, Buerger's disease, multiple sclerosis and type I diabetes);
6. Concomitant malignancy or previous malignancy within 5 years before enrolment, excluding skin cancer, local prostate cancer or cervical carcinoma in situ;
7. Organ transplant recipients;
8. Patients with active auto-immune disorder, e.g. autoimmune hepatitis, systemic lupus erythematous etc.;
9. Severe dysfunction of the heart, kidney, or other organs;
10. Severe psychological dysfunction;
11. Sensitive to cytokines, any reagent or associated component in MASCT;
12. Ever participated in any clinical trial of other drugs within 3 months before enrolment;
13. Other patients that investigators think unsuitable to be enrolled.

Inclusion Criteria before immunotherapy:

1. Imaging (enhanced CT or MRI) confirmed completely tumor necrosis or tumor removed 4 weeks after RFA/Hepatectomy；
2. Obtaining adequate samples of the matched tumor and adjacent nontumor normal liver tissues;
3. Sensitive mutations can be detected by gene sequencing in tumour tissue;
4. Prediction of neoantigen peptides ≥10;
5. Synthesized neo antigen peptides ≥5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2-year
  Defined in whole days as the time from randomisation until disease recurrence or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and relapse free. Patients not having an event will be censored at the date last seen alive and relapse free.
Immune response rate | 2-year
  The demonstration of immune response is potentially related to prognosis and will be quantified in both groups because ablative therapy alone has been shown to induce anti-tumour immune responses.

SECONDARY OUTCOMES:
Overall survival | 2-year
  Defined in whole days as the time from randomisation until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.
Recurrence rate | 2-year
  The rate of HCC recurrence in the total number of patients.
Safety events | 2-year
  Safety events will be measured in terms of the occurrence, severity, type and causality of Adverse Events (AEs) during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 4).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991
- [Background] Ali MY, Grimm CF, Ritter M, Mohr L, Allgaier HP, Weth R, Bocher WO, Endrulat K, Blum HE, Geissler M. Activation of dendritic cells by local ablation of hepatocellular carcinoma. J Hepatol. 2005 Nov;43(5):817-22. doi: 10.1016/j.jhep.2005.04.016. Epub 2005 Jun 20. PMID 16087270
- [Background] Shi L, Chen L, Wu C, Zhu Y, Xu B, Zheng X, Sun M, Wen W, Dai X, Yang M, Lv Q, Lu B, Jiang J. PD-1 Blockade Boosts Radiofrequency Ablation-Elicited Adaptive Immune Responses against Tumor. Clin Cancer Res. 2016 Mar 1;22(5):1173-1184. doi: 10.1158/1078-0432.CCR-15-1352. PMID 26933175
- [Background] Wissniowski TT, Hansler J, Neureiter D, Frieser M, Schaber S, Esslinger B, Voll R, Strobel D, Hahn EG, Schuppan D. Activation of tumor-specific T lymphocytes by radio-frequency ablation of the VX2 hepatoma in rabbits. Cancer Res. 2003 Oct 1;63(19):6496-500. PMID 14559842
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Derived] Peng S, Chen S, Hu W, Mei J, Zeng X, Su T, Wang W, Chen Z, Xiao H, Zhou Q, Li B, Xie Y, Hu H, He M, Han Y, Tang L, Ma Y, Li X, Zhou X, Dai Z, Liu Z, Tan J, Xu L, Li S, Shen S, Li D, Lai J, Peng B, Peng Z, Kuang M. Combination Neoantigen-Based Dendritic Cell Vaccination and Adoptive T-Cell Transfer Induces Antitumor Responses Against Recurrence of Hepatocellular Carcinoma. Cancer Immunol Res. 2022 Jun 3;10(6):728-744. doi: 10.1158/2326-6066.CIR-21-0931. PMID 35476700